CLINICAL TRIAL: NCT00105508
Title: A Double-blind, Placebo-controlled, Multicenter, Multinational Phase III Study to Evaluate the Safety and Efficacy of Sarizotan HCl 1 mg b.i.d. in Patients With Parkinson's Disease Suffering From Treatment-associated Dyskinesia
Brief Title: Sarizotan HC1 in Patients With Parkinson's Disease Suffering From Treatment-associated Dyskinesia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR 62225-018
Record Dates: First submitted 2005-03-15; First posted 2005-03-16 (Estimated); Results first posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Parkinson's Disease; Dyskinesia
Keywords: Parkinson's Disease; Dyskinesia; Dyskinesia associated with dopaminergic treatment
MeSH Terms: conditions — Parkinson Disease; Dyskinesias | interventions — sarizotan

ARMS (2):
- Sarizotan (Experimental)
  Interventions: Drug: Sarizotan
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sarizotan — Subjects will receive sarizotan 1 milligram orally twice daily for 24 weeks.
  Arms: Sarizotan
Drug: Placebo — Subjects will receive placebo matched to sarizotan orally twice daily for 24 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if Sarizotan HC1 1 mg b.i.d. (taken twice a day) is effective in the treatment of dyskinesia associated with dopaminergic treatment of Parkinson's disease (PD).

ELIGIBILITY:
Inclusion Criteria:

* The subject is an out-patient.
* The subject presents with a diagnosis of idiopathic Parkinson's disease.
* Prior therapy with all registered Parkinsonian medication is allowed.

Exclusion Criteria:

* (For female subjects) The subject is pregnant or lactating.
* The subject is participating in another clinical study or has done so within the past 30 days.
* The subject has received neurosurgical intervention related to PD.
* The subject has relevant renal impairment.
* The subject has relevant hepatic impairment.
* The subject is suffering from any dementia or psychiatric illness.
* The subject has a history of allergic asthma.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 506 (Actual)
Dates: Start 2004-09-30 (Actual); Primary Completion 2006-02-28 (Actual); Study Completion 2006-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Inc., a business of Merck KGaA, Darmstadt, Germany
Locations (29):
- United States (29):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - La Jolla, California
  - Oxnard, California
  - Sacramento, California
  - Englewood, Colorado
  - Danbury, Connecticut
  - Farmington, Connecticut
  - Jacksonville, Florida
  - Maitland, Florida
  - St. Petersburg, Florida
  - Decatur, Georgia
  - Chicago, Illinois
  - Springfield, Illinois
  - Des Moines, Iowa
  - New Orleans, Louisiana
  - Scarborough, Maine
  - Boston, Massachusetts
  - Southfield, Michigan
  - Edison, New Jersey
  - New Hyde Park, New York
  - New York, New York
  - Durham, North Carolina
  - Oklahoma City, Oklahoma
  - Pittsburgh, Pennsylvania
  - Brentwood, Tennessee
  - South Ogden, Utah
  - Spokane, Washington
  - Milwaukee, Wisconsin

REFERENCES:
- [Result] Goetz CG, Laska E, Hicking C, Damier P, Muller T, Nutt J, Warren Olanow C, Rascol O, Russ H. Placebo influences on dyskinesia in Parkinson's disease. Mov Disord. 2008 Apr 15;23(5):700-7. doi: 10.1002/mds.21897. PMID 18175337
- See also: EudraCT results summary synopsis — https://www.clinicaltrialsregister.eu/ctr-search/trial/2004-001593-10/results

RESULTS

PARTICIPANT FLOW:
Groups:
- Sarizotan: Subjects received sarizotan 1 milligram orally twice daily for 24 weeks.
- Placebo: Subjects received placebo matched to sarizotan orally twice daily for 24 weeks.
Period: Overall Study
Arm/Group | Sarizotan | Placebo
Started | 253 | 253
Completed | 213 | 217
Not Completed | 40 | 36
Not completed — Prephase Dropout | 1 | 0
Not completed — Adverse Event | 16 | 19
Not completed — Insufficient Efficacy | 1 | 0
Not completed — Withdrawal by Subject | 10 | 6
Not completed — Lost to Follow-up | 3 | 0
Not completed — Protocol Violation | 1 | 2
Not completed — Other | 8 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sarizotan | Placebo | Total
Number analyzed (Participants) | 253 | 253 | 506
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (9.93) | 65.0 (9.11) | 64.1 (9.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126 | 112 | 238
  Male | 127 | 141 | 268

OUTCOME MEASURES:

1. Primary Outcome: Responder Rate Based on Unified Parkinson's Disease Rating Scale (UPDRS) Items 32 and 33 at Week 12
Description: Responder rate was defined as the percentage of subjects with 25% improvement compared to baseline in the sum of UPDRS scores for items 32 and 33. The UPDRS was an investigator-assessed rating tool to follow the longitudinal course of Parkinson's disease. Items 32 and 33 assessed duration of dyskinesia and disability due to dyskinesia, respectively. Both items were rated on a 0 to 4-point scale, where higher scores indicated higher duration of dyskinesia and more disability due to dyskinesia, respectively. The Items 32 and 33 composite score was sum of the individual item scores and ranged from 0 to 8, where higher score indicated more complications due to dyskinesia.
Time Frame: Week 12
Population: Intent to treat population included all subjects who were randomized in the study.
Measure: Number; unit: percentage of subjects
Arm/Group | Sarizotan | Placebo
Number analyzed (Participants) | 253 | 253
percentage of subjects | 30.4 | 33.2

2. Primary Outcome: Responder Rate Based on Unified Parkinson's Disease Rating Scale (UPDRS) Items 32 and 33 at Week 24
Description: as for outcome 1
Time Frame: Week 24
Population: Intent to treat population included all subjects who were randomized in the study.
Measure: Number; unit: percentage of subjects
Arm/Group | Sarizotan | Placebo
Number analyzed (Participants) | 253 | 253
percentage of subjects | 37.2 | 39.5

3. Primary Outcome: Change From Baseline in Unified Parkinson's Disease Rating Scale (UPDRS) Total Score for Items 18 to 31 at Week 12
Description: The UPDRS was an investigator-assessed rating tool to follow the longitudinal course of Parkinson's disease. Each item from 18 to 31 was rated on a scale ranging from 0 to 4, where higher scores indicated higher complications due to dyskinesia. The total score was the sum of the individual item scores and ranged from 0 to 56, where higher score indicated more complications due to dyskinesia. Change = Week 12 - Baseline.
Time Frame: Baseline, Week 12
Population: Intent to treat population included all subjects who were randomized in the study. Here "Overall Number of Participants Analyzed" signifies those subjects who were evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sarizotan | Placebo
Number analyzed (Participants) | 253 | 251
units on a scale | 0.1 (7.45) | -0.2 (0.0)

4. Primary Outcome: Change From Baseline in Unified Parkinson's Disease Rating Scale (UPDRS) Total Score for Items 18 to 31 at Week 24
Description: The UPDRS was an investigator-assessed rating tool to follow the longitudinal course of Parkinson's disease. Each item from 18 to 31 was rated on a scale ranging from 0 to 4, where higher scores indicated higher complications due to dyskinesia. The total score was the sum of the individual item scores and ranged from 0 to 56, where higher score indicated more complications due to dyskinesia. Change = Week 24 - Baseline.
Time Frame: Baseline, Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sarizotan | Placebo
Number analyzed (Participants) | 253 | 251
units on a scale | -0.2 (7.92) | -0.0 (6.61)

ADVERSE EVENTS:
Description: Safety population was used for adverse events. Safety population included those subjects who received at least 1 dose of study drug or placebo.
Arm/Group | Sarizotan | Placebo
Serious Adverse Events (participants affected / at risk) | 23/252 | 25/252
Other Adverse Events (participants affected / at risk) | 100/252 | 86/252
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sarizotan (N=252) | Placebo (N=252)
Fall (Injury, poisoning and procedural complications) | 1 | 3
Hepatic trauma (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Dyskinesia (Nervous system disorders) | 1 | 1
Dystonia (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1
Parkinsonism (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 1 | 1
Abscess limb (Infections and infestations) | 0 | 1
Arthritis bacterial (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 3
Urosepsis (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 1 | 0
Hernia repair (Surgical and medical procedures) | 1 | 0
Hip arthroplasty (Surgical and medical procedures) | 0 | 1
Hip surgery (Surgical and medical procedures) | 0 | 1
Knee arthroplasty (Surgical and medical procedures) | 1 | 0
Spinal fusion surgery (Surgical and medical procedures) | 1 | 0
Spinal nerve stimulator implantation (Surgical and medical procedures) | 1 | 0
Surgery (Surgical and medical procedures) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 1 | 1
Crohn's disease (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Electrocardiogram change (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Investigation (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Coronary artery insufficiency (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Nodal arrhythmia (Cardiac disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 1
Asthenia (General disorders) | 1 | 0
Local swelling (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sarizotan (N=252) | Placebo (N=252)
Dyskinesia (Nervous system disorders) | 24 | 19
Parkinsonism (Nervous system disorders) | 24 | 24
Fall (Injury, poisoning and procedural complications) | 28 | 21
Depression (Psychiatric disorders) | 15 | 7
Nausea (Gastrointestinal disorders) | 9 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other